CLINICAL TRIAL: NCT07083973
Title: Prone Position Assessment by 3D EIT in ARDS Patients
Brief Title: Prone Position Assessed by 3D EIT
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Prone position by 3D-EIT
Record Dates: First submitted 2024-11-14; First posted 2025-07-24 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome); Respiratory Failure
MeSH Terms: conditions — Acute Lung Injury; Respiratory Insufficiency | interventions — Prone Position

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Prone position — Patients were ventilated based on the ARDS-Net recommendations . Patients were kept in a supine position. The process of lung ventilation and perfusion assessment was as follows:
  1. PEEP was determined by the attending doctor and was kept the same during the supine and prone period.
  2. 3D-EIT was used to monitor the ventilation and perfusion of ARDS patients at three timepoints: T1: supine position, T2: prone position at 30min, T3: prone position over 10 hours.

SUMMARY:
To investigate global and regional changes in lung ventilation and perfusion induced by prone position in ARDS patients assessed by 3D-EIT. And to investigate the difference between 2D-EIT and 3D-EIT in prone position monitoring.

ELIGIBILITY:
Inclusion Criteria:

* patients on mechanical ventilation.
* Diagnosis of ARDS was based on the Berlin definition
* Patients in need of prone position because of clinical condition

Exclusion Criteria:

* Under 18 years of age.
* Pregnant women;
* Ribcage malformation
* Any contraindication to the use of EIT (e.g. automatic implantable cardioverter defibrillator, and implantable pumps).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ARDS on mechanical ventilation
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Regional ventilation monitored by EIT | 5-10minutes
  Using EIT to monitor the regional ventilation during supine and prone position, to monitor the ventilation distribution change.
Regional perfusion monitored by EIT | 5-10minutes
  Using EIT to monitor the regional perfusion during supine and prone position, to monitor the ventilation distribution change.
V/Q monitored by EIT | 5-10minutes
  Ventilation and perfusion monitored by EIT in supine and prone position. To evaluate the V/Q match, deadspace and shunt lung region.

SECONDARY OUTCOMES:
Respiratory system compliance | 1 day
  Monitor the respiratory system compliance during supine and prone position
SpO2 | 1 day
  Monitor the SpO2 during supine and prone position

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine, Peking Union Medical College Hospital, Peking Union Medical College, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China